CLINICAL TRIAL: NCT04841915
Title: A Randomized Controlled Trial of Effects of DAIry PROtein Products on Liver Disease Severity and Metabolism in Patients With Non-Alcoholic Fatty Liver Disease.
Brief Title: Dairy Protien Rich Diet for NAFLD Patients
Acronym: DAIPRO-NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry); University of Copenhagen (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIPRO-NAFLD
Record Dates: First submitted 2021-03-24; First posted 2021-04-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2023-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Metabolic Syndrome; Caseins; Whey; Diet, High Protein; Weight Loss; Lipoproteins, VLDL
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Weight Loss | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants will be randomized to one of 3 treatment arms. Protein interventions (MCI and WPI) will be blinded to participants and investigators, but controls with regular diet will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Micellar Cassein Isolate High-Protein Diet (Experimental): 4weeks eucaloric intake on high-protein diet with micellar cassein as primary protein source followed by 20weeks hypocaloric intake on equivalent protein rich diet.
  Interventions: Dietary Supplement: High-Protein Diet; Behavioral: Clinical dietician; Behavioral: Weight loss
- Whey Protein High-Protein Diet (Experimental): 4weeks eucaloric intake on high-protein diet with whey protein as primary protein source followed by 20weeks hypocaloric intake on equivalent protein rich diet.
  Interventions: Dietary Supplement: High-Protein Diet; Behavioral: Clinical dietician; Behavioral: Weight loss
- Normal Diet (Placebo Comparator): 4weeks eucaloric diet with normal protein content (15E%) followed by 20weeks hypocaloric intake on equivalent diet.
  Interventions: Behavioral: Clinical dietician; Behavioral: Weight loss

INTERVENTIONS:
Dietary Supplement: High-Protein Diet — Diet consisting of 25E% from assigned protein during eucaloric diet and 35E% from assigned protein during hypocaloric diet
  Arms: Micellar Cassein Isolate High-Protein Diet; Whey Protein High-Protein Diet
Behavioral: Clinical dietician — Counselling from a clinical dietician bi-weekly until weight loss of 5% is achieved.
Behavioral: Weight loss — 4 weeks eucaloric diet ~13 MJ/day followed by, 20 weeks hypocaloric diet ~9 MJ/day until 5% weight loss is achieved.

SUMMARY:
The overarching aim of this project is to investigate effects of dietary interventions on nonalcoholic fatty liver disease (NAFLD) severity and to delineate the relationship with improvements in metabolic aberrations in liver-, fat- and muscle tissue, using a panel of state-of-the art techniques.

The investigators will conduct a randomized clinical trial with three arms to investigate if micellar cassein isolate and whey protein supplementation as part of a high-protein diet during 4 weeks of weight maintenance and 20 weeks of hypocaloric intake (30% energy restriction) inducing modest weight loss (5% of baseline weight) has beneficial effects on NAFLD severity and metabolic aberrations compared to normal diet in NAFLD patients.

It is hypothesized that: (i) a high-protein diet improves liver disease severity and metabolic function compared to a normal protein diet; (ii) Cassein provides greater benefits than whey; and(iii) these effects manifest during both weight maintenance and weight loss.

DETAILED DESCRIPTION:
To test the hypothesis, state-of-the-art techniques for a comprehensive assessment of liver disease severity and metabolic function will be employed. NAFLD severity and treatment effects will be evaluated on the basis of liver fat content (MR spectroscopy), liver enzymes, liver-specific inflammation and fibrosis markers and fibrosis (fibroscan). Metabolic function will be investigated by basal and insulin mediated whole-body glucose, fatty acid and VLDL-TG turnover, postprandial insulin secretion and clearance (mixed meal test in conjunction with oral minimal modeling). Body composition (total fat mass, leg fat and fat free mass) will be assessed by DEXA-scanning; visceral and upper-body subcutaneous fat by MR-imaging, and fat content of skeletal muscle and liver by MR-spectroscopy. All outcomes will be assessed at baseline, after 4 wk on a eucaloric diet (weight maintenance), and after an additional 20 wk on a hypocaloric diet (5% weight loss), in 54 patients with NAFLD and obesity (BMI ≥30 kg/m2) but without diabetes. Subjects will be block randomized to one of three treatment groups (WPI, MCI, or standard diet, n=18 in each group). A biobank of serum/plasma/DNA including fat and skeletal muscle biopsies will be established for mechanistic analysis in a planned future work-package. Patient related outcomes will include specific questionnaires (CLDQ-NAFLD, SF-36).

All subjects will be phone-contacted on a regular basis by study personnel to monitor progress, resolve problems with the diets, and reinforce compliance; and meet in person with the study dietitians weekly during the weight maintenance phase and biweekly during the weight loss phase to have their body weight measured and receive dietary counselling. Before study initiation, the research teams will put together standardized procedures for patient contact and nutrition counselling, including creating nutrition information leaflets specific to each randomization arm, to ensure uniformity between the study centers. In practice, dietary guidance will be tailored to the individual patient to ensure weight maintenance within 2% of baseline body weight during the first phase (weight stability), and a weight loss of 0.25% per week to reach the target 5% weight loss after 20 weeks during the second phase (weight loss); energy intake will be adjusted as necessary by adding or removing carbohydrate to meet the desired goals. Three-day diet records will be collected before and every 2 weeks during the interventions to evaluate energy and macronutrient intakes. A 3-hour urine sample will be collected during the mixed meal test at baseline, after 4 and 24 weeks in order to monitor dietary protein intake. Participants will be instructed in how to do the sampling and storing the sample cool during the collection.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27.5 kg/m2
* HbA1C < 48 mmol/mol
* Written informed consent
* Liver steatosis > 10% on MR-spectroscopy
* Premenopausal women will have a negative pregnancy test drawn within 48 hours before the study.

Exclusion Criteria:

* Other chronic liver diseases (HBV, HCV, AIH, PBC, PSC, alcoholic steatosis)
* Known systemic disease exempting hypertension and dyslipidemia.
* Former or active malignant disease
* Alcohol consumption >2 drinks/day for men, 1 drink/day for women, evaluated by AUDIT-C
* Pregnancy
* Any medications including non-prescription medications exempting, birth control medications, antihypertensives and statins. Participants taking statins can participate on the condition of a 2 week pause before the experimental days.
* Estimated glomerular filtration rate <90 ml/min
* Currently smoking
* Blood donation within the last 3 months
* Weight above 130 kg
* Participated in trials using radioactive isotopes within the last 6 months

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Steatosis, absolute | 4 weeks and 20 weeks
  Absolute difference in changes in steatosis (MRs) between diets
Steatosis, relative | 4 weeks and 20 weeks
  Relative difference in changes in steatosis (MRs) between diets
Liver enzymes | 4 weeks and 20 weeks
  Difference in change of liver enzymes between diets

SECONDARY OUTCOMES:
Hepatic Insulin Resistance | 24 weeks
  Changes in hepatic insulin resistance measured by changes in suppression of EGP from basal period to clamp period.
Adipose tissue Insulin Resistance | 24 weeks
  Changes in adipose insulin resistance measured by changes in suppression of lipolysis from basal period to clamp period.
Peripheral insulin resistance | 24 weeks
  Changes in peripheral insulin resistance measured total rate of disappearance of glucose in hyperinsulinemic clamp.
Insulin Secretion | 24 weeks
  Changes in Insulin Secretion

OTHER OUTCOMES:
Anthropometric measures | 24 weeks
  Changes in body composition (Fat mass, lean mass, waist-hip-ratio, BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Prof., Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Dept. Hepatology and Gastroenterology, Aarhus N
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No